CLINICAL TRIAL: NCT03792841
Title: A Phase 1 Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Efficacy of Prostate Specific Membrane Antigen Half-life Extended Bispecific T-cell Engager Acapatamab in Subjects With Metastatic Castration-resistant Prostate Cancer
Brief Title: Safety, Tolerability, Pharmacokinetics, and Efficacy of Acapatamab in Subjects With mCRPC
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20180101
Record Dates: First submitted 2019-01-02; First posted 2019-01-03 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Metastatic Castration-resistant Prostate Cancer; Prostate Cancer
Keywords: acapatamab; HLE-BiTE®; mCRPC; Metastatic Castration-resistant Prostate Cancer; Prostate cancer; PSMA; BiTE®; Bispecific T-Cell engager; Immunotherapy; Immuno-oncology; Immunooncology; Solid tumor; PSMA Targeted Therapy
MeSH Terms: conditions — Prostatic Neoplasms; Bites and Stings | interventions — pembrolizumab; Immune Checkpoint Inhibitors; Etanercept; Cytochrome P-450 Enzyme System

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Part 1 Dose-exploration: acapatamab treatment (Experimental): Part 1 dose-exploration: acapatamab is administered intravenously. The dose-exploration phase of the study will estimate the MTD of acapatamab. RP2D may be identified based on emerging safety, efficacy, and pharmacodynamic data prior to reaching an MTD.
  Interventions: Drug: acapatamab
- Part 1 Dose-expansion: acapatamab treatment (Experimental): Part 1 dose-expansion: acapatamab is administered intravenously at the MTD/RP2D.
  Interventions: Drug: acapatamab
- Part 2: acapatamab + Pembrolizumab (Experimental): Part 2: acapatamab is administered intravenously at the MTD/RP2D. Pembrolizumab will be administered intravenously.
  Interventions: Drug: acapatamab; Drug: Pembrolizumab
- Part 3: acapatamab + Etanercept Prophylaxis (Experimental): Part 3: acapatamab is administered intravenously at RP2D/MTD levels. Etanercept will be administered subcutaneously in cycle 1 only.
  Interventions: Drug: acapatamab; Drug: Etanercept
- Part 4: acapatamab 24 Hour Monitoring (Experimental): Part 4: acapatamab is administered intravenously at RP2D/MTD with 24-hour monitoring.
  Interventions: Drug: acapatamab
- Part 5: acapatamab Outpatient Cohort (Experimental): Part 5: acapatamab is administered intravenously at RP2D/MTD in an outpatient setting with 8-hour monitoring.
  Interventions: Drug: acapatamab
- Part 6: acapatamab + Cytochrome P450 (CYP) Cocktail Drug Interaction (Experimental): Part 6: acapatamab is administered intravenously at RP2D/MTD. A CYP phenotyping cocktail will be administered orally.
  Interventions: Drug: acapatamab; Drug: Cytochrome P450 (CYP) Cocktail

INTERVENTIONS:
Drug: acapatamab — Investigational immunotherapy for the treatment of metastatic castration-resistant prostate cancer
  Other Names: PSMA Targeted Therapy
Drug: Pembrolizumab — Combined with acapatamab for investigational treatment of mCRPC
  Other Names: PD-1 inhibitor
  Arms: Part 2: acapatamab + Pembrolizumab
Drug: Etanercept — Prophylaxis for acapatamab-related cytokine release syndrome.
  Other Names: TNF-alpha inhibitor
  Arms: Part 3: acapatamab + Etanercept Prophylaxis
Drug: Cytochrome P450 (CYP) Cocktail — Evaluate the effect of co-administration of multiple dosing of acapatamab on plasma
  Other Names: Cooperstown 5+1 CYP phenotyping cocktail
  Arms: Part 6: acapatamab + Cytochrome P450 (CYP) Cocktail Drug Interaction

SUMMARY:
A phase 1 study evaluating the safety, tolerability, pharmacokinetics, and efficacy of prostate specific membrane antigen half-life extended bispecific T-cell engager acapatamab in subjects with metastatic castration-resistant prostate cancer, and to determine the maximum tolerated dose (MTD) or recommended phase 2 dose (RP2D).

DETAILED DESCRIPTION:
This is a phase I, first-in-human study to evaluate the safety and tolerability of acapatamab; a half-life extended (HLE) bispecific T-cell engager (BiTE®) construct, alone and in combination with pembrolizumab, etanercept prophylaxis and cytochrome P450 (CYP) phenotyping cocktail in subjects with metastatic castration-resistant prostate cancer.

ELIGIBILITY:
All Parts

Inclusion Criteria:

* Subject has provided informed consent prior to initiation of any study specific activities/procedures
* Subjects with histologically or cytologically confirmed mCRPC who are refractory to a novel antiandrogen therapy (abiraterone, enzalutamide, and/or apalutamide) and have failed at least 1 (but not more than 2) taxane regimens (or who are deemed medically unsuitable to be treated with a taxane regimen or have actively refused treatment with a taxane regimen). Progression on novel antiandrogen therapy may have occurred in the non-metastatic CRPC setting
* Subjects must have undergone bilateral orchiectomy or must be on continuous ADT with a gonadotropin releasing hormone (GnRH) agonist or antagonist
* Total serum testosterone </= 50 ng/dL or 1.7 nmol/L
* Evidence of progressive disease, defined as 1 or more PCWG3 criteria:
* PSA level >/= 1 ng/mL that has increased on at least 2 successive occasions at least 1 week apart
* nodal or visceral progression as defined by RECIST 1.1 with PCGW3 modifications
* appearance of 2 or more new lesions in bone scan
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 1
* Life expectancy >/= 6months

Exclusion Criteria:

* Any anticancer therapy or immunotherapy within 4 weeks of start of first dose, not including luteinizing hormone-releasing hormone agonist (LHRH)/GnRH analogue (agonist/antagonist). Subjects on a stable bisophosphonate or denosumab regimen for >/= 30 days prior to randomization are eligible
* Prior PSMA-targeted therapy (subjects on prior therapy may be eligible if discussed with Amgen medical monitor prior to enrollment)
* Central nervous system (CNS) metastases, leptomeningeal disease, or spinal cord compression
* Active autoimmune disease or any other diseases requiring immunosuppressive therapy while on study
* Needing chronic systemic corticosteroid therapy (prednisone > 10 mg per day or equivalent) or any other immunosuppressive therapies (including anti-tumor necrosis factor alpha [TNF alpha] therapies) unless stopped 7 days prior to start of first dose
* Myocardial infarction, unstable angina, cardiac arrhythmia requiring medication, and/or symptomatic congestive heart failure (New York Heart Association > class II) within 12 months of first dose of acapatamab

Part 2 only:

* Subjects on a prior PD-1 or PD-L1 inhibitor who experienced a Grade 3 or higher immune-related adverse event prior to first day of dosing
* History or evidence of interstitial lung disease or active, non-infectious pneumonitis

Part 3 only:

- Evidence of active tuberculosis on chest radiograph within 3 months prior to the first dose of investigational product

Part 6 only:

Subjects are excluded from this cohort if any of the following additional criteria apply:

* Subjects taking strong OAT3 inhibitors (eg, probenecid) or adjust the dosing to 1 mg PO QD.
* Subjects with latent or active tuberculosis at screening

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2019-02-05 (Actual); Primary Completion 2023-06-29 (Actual); Study Completion 2023-06-29 (Actual)

PRIMARY OUTCOMES:
Number of participants with dose-limiting toxicity | Up to 3 years
  Parts 1, 2, 3, 4, 5, and 6 of the study
Number of participants with treatment-emergent adverse events | Up to 3 years
  Parts 1, 2, 3, 4, 5, and 6 of the study
Number of participants with treatment-related adverse events | Up to 3 years
  Parts 1, 2, 3, 4, 5, and 6 of the study
Number of participants with clinically significant changes in vital signs | Up to 3 years
  Parts 1, 2, 3, 4, 5, and 6 of the study
Number of participants with clinically significant changes in electrocardiogram (ECG) | Up to 3 years
  Parts 1, 2, 3, 4, 5, and 6 of the study
Number of participants with clinically significant changes in clinical laboratory tests | Up to 3 years
  Parts 1, 2, 3, 4, 5, and 6 of the study

SECONDARY OUTCOMES:
Maximum serum concentration (Cmax) of acapatamab | Up to 3 years
  Parts 1, 2, 3, 4, 5, and 6 of the study
Minimum serum concentration (Cmin) of acapatamab | Up to 3 years
  Parts 1, 2, 3, 4, 5, and 6 of the study
Area under the concentration-time curve (AUC) over the dosing interval of acapatamab | Up to 3 years
  Parts 1, 2, 3, 4, 5, and 6 of the study
Accumulation ratio of acapatamab | Up to 3 years
  Parts 1, 2, 3, 4, 5, and 6 of the study
Half-life of acapatamab | Up to 3 years
  Parts 1, 2, 3, 4, 5, and 6 of the study
Objective response (OR) | Up to 3 years
  Parts 1, 2, 3, 4, 5, and 6 of the study
Prostate-specific antigen (PSA) response | Up to 3 years
  Parts 1, 2, 3, 4, 5, and 6 of the study
Duration of response (DOR) (radiographic and PSA) | Up to 3 years
  Parts 1, 2, 3, 4, 5, and 6 of the study
Percentage of participants experiencing a response based on 68Gallium (68Ga)-prostate-specific membrane antigen (PSMA)-11 positron emission tomography (PET)/computed tomography (CT) response evaluations | Up to 3 years
  Parts 1, 2 and 3 only.
Percentage of participants experiencing a response based on 18F-fluorodeoxyglucose (FDG) positron emission tomography (PET)/computed tomography (CT) response evaluations | Up to 3 years
  Parts 1, 2 and 3 only.
Change in time to progression (radiographic and PSA) | Up to 3 years
  Parts 1, 2, 3, 4, 5, and 6 of the study
Progression-free survival (PFS) (radiographic and PSA) | Up to 3 years
  Parts 1, 2, 3, 4, 5, and 6 of the study.
1, 2 and 3-year overall survival (OS) | Up to 3 years
  Parts 1, 2, 3, 4, 5, and 6 of the study
Percentage of participants experiencing circulating tumor cells (CTC) response | Up to 3 years
  Parts 1, 2, 3, 4, 5, and 6 of the study. CTC response defined as CTC0 (reduction of CTCs > 0 to 0) or CTC conversion (≥ 5 CTCs/7.5 mL blood to ≤ 4 CTCs/7.5 mL blood)
Other PCWG3-recommended endpoints - time to symptomatic skeletal events | Up to 3 years
  Parts 1, 2, 3, 4, 5, and 6 of the study
Other PCWG3-recommended endpoints - lactate dehydrogenase [LDH] levels | Up to 3 years
  Parts 1, 2, 3, 4, 5, and 6 of the study
Other PCWG3-recommended endpoints - hemoglobin levels | Up to 3 years
  Parts 1, 2, 3, 4, 5, and 6 of the study
Other PCWG3-recommended endpoints - neutrophil-to-lymphocyte ratio | Up to 3 years
  Parts 1, 2, 3, 4, 5, and 6 of the study
Other PCWG3-recommended endpoints - urine N-telopeptide levels | Up to 3 years
  Parts 1, 2, 3, 4, 5, and 6 of the study
Other PCWG3-recommended endpoints - alkaline phosphatase [total, bone] levels | Up to 3 years
  Parts 1, 2, 3, 4, 5, and 6 of the study
Maximum serum concentration (Cmax) of acapatamab when administered with CYP enzymes | Up to 3 years
  Part 6 only.
Area under the concentration-time curve over a 24-hour period (AUC24) of acapatamab when administered with CYP enzymes | Up to 3 years
  Part 6 only.
Half-life of acapatamab when administered with CYP enzymes | Up to 3 years
  Part 6 only.

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (30):
- United States (13):
  - El Camino Hospital, Campbell, California
  - City of Hope National Medical Center, Duarte, California
  - City of Hope at Long Beach Elm, Long Beach, California
  - University of California Los Angeles, Los Angeles, California
  - Emory University, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Tulane Medical Center, New Orleans, Louisiana
  - Washington University, St Louis, Missouri
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Cornell Medical College, New York, New York
  - University of Texas Southwestern Medical Center, Dallas, Texas
- Australia (3):
  - Chris OBrien Lifehouse, Camperdown, New South Wales
  - Scientia Clinical Research Ltd, Randwick, New South Wales
  - Peter MacCallum Cancer Centre, Parkville, Victoria
- Austria (4):
  - Ordensklinikum Linz Elisabethinen, Linz
  - Landeskrankenhaus Salzburg, Salzburg
  - Krankenhaus der Barmherzigen Brueder Wien, Vienna
  - Universitaetsklinikum Allgemeines Krankenhaus Wien, Vienna
- Belgium (2):
  - Universite Catholique de Louvain Cliniques Universitaires Saint Luc, Brussels
  - Universitair Ziekenhuis Gent, Ghent
- BC Cancer Vancouver, Vancouver, British Columbia, Canada
- Institut Gustave Roussy, Villejuif, France
- Japan (2):
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - Yokohama City University Medical Center, Yokohama, Kanagawa
- Erasmus Medisch Centrum, Rotterdam, Netherlands
- Singapore (2):
  - National University Hospital, Singapore
  - National Cancer Centre Singapore, Singapore
- Linkou Chang Gung Memorial Hospital of Chang Gung Medical Foundation, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe, or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Background] Dorff T, Horvath LG, Autio K, Bernard-Tessier A, Rettig MB, Machiels JP, Bilen MA, Lolkema MP, Adra N, Rottey S, Greil R, Matsubara N, Tan DSW, Wong A, Uemura H, Lemech C, Meran J, Yu Y, Minocha M, McComb M, Penny HL, Gupta V, Hu X, Jurida G, Kouros-Mehr H, Janat-Amsbury MM, Eggert T, Tran B. A Phase I Study of Acapatamab, a Half-life Extended, PSMA-Targeting Bispecific T-cell Engager for Metastatic Castration-Resistant Prostate Cancer. Clin Cancer Res. 2024 Apr 15;30(8):1488-1500. doi: 10.1158/1078-0432.CCR-23-2978. PMID 38300720
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com